CLINICAL TRIAL: NCT06311942
Title: Effectiveness of Triple Versus Dual Adjuvant Therapy in VETC-positive Population Following Liver Resection for HCC: a Prospective Multicenter Cohort Study
Brief Title: Triple vs. Dual Adjuvant Therapy Following Liver Resection for HCC.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Precision AT-02
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: HCC
Keywords: HCC; Adjuvant therapy; VETC; HAIC; Lenvatinib; PD-1 inhibitors
MeSH Terms: interventions — Immune Checkpoint Inhibitors; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple adjuvant therapy group (Experimental): Patients in the triple adjuvant therapy group received HAIC in combination with PD-1 inhibitors and lenvatinib adjuvant therapy.
  Interventions: Drug: HAIC plus PD-1 inhibitors plus lenvatinib
- Dual adjuvant therapy group (Active Comparator): Patients in the Dual adjuvant therapy group received PD-1 inhibitors combined lenvatinib adjuvant therapy.
  Interventions: Drug: PD-1 inhibitors plus lenvatinib

INTERVENTIONS:
Drug: HAIC plus PD-1 inhibitors plus lenvatinib — Patients in the triple adjuvant therapy group received one cycle of HAIC about a month after liver resection, HAIC was adopted the FOFOLX6 program (Folinic acid+5-fluorouracil+Oxaliplatin). The first cycle of PD-1 monoclonal antibody was administrated 2-4 weeks postoperatively, 200 mg IV, every 21 days for a total of 9 cycles. Lenvatinib was initiated orally 2-4 weeks postoperatively for 6 months.
  Other Names: Non
  Arms: Triple adjuvant therapy group
Drug: PD-1 inhibitors plus lenvatinib — The first cycle of PD-1 monoclonal antibody was administrated 2-4 weeks postoperatively, 200 mg IV, every 21 days for a total of 9 cycles. Lenvatinib was initiated orally 2-4 weeks postoperatively for 6 months.
  Other Names: Non
  Arms: Dual adjuvant therapy group

SUMMARY:
Vessels that encapsulate tumor clusters (VETC) is an invasive metastatic factor in HCC independent of the epithelial mesenchyme transition (EMT), and VETC-positive patients have a higher rate of postoperative recurrence. What can be done to improve the surgical prognosis of this group of patients needs to be continuously explored.

DETAILED DESCRIPTION:
Previous studies have identified VETC as a new metastatic pattern independent of EMT that may be associated with immunosuppression as well as poor prognosis. Multiple retrospective studies find higher rates of postoperative recurrence, distant metastasis in VETC-positive patients. How to improve surgical prognosis in VETC-positive patients needs to be explored. In recent years, adjuvant immunotherapy (sintilimab) and adjuvant immunotherapy combined with targeted therapy (T+A) have been shown to be effective in improving the surgical prognosis. There are no published studies on how to improve prognosis for VETC-positive population. One of our unpublished retrospective studies found that VETC-positive patients receiving PD-1 monoclonal antibody was not effective in improving prognosis, however, PD-1 inhibitor combined with lenvatinib reduces recurrences significantly. In addition, some studies have also found that postoperative adjuvant hepatic artery infusion chemotherapy (HAIC) is also potentially useful in improving surgical prognosis. It is not clear whether triple therapy can further reduce recurrence in these tumors, which have highly aggressive characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75.
2. No previous local or systemic treatment for hepatocellular carcinoma.
3. Child-Pugh liver function score ≤ 7.
4. ECOG PS 0-1.
5. No serious organic diseases of the heart, lungs, brain, kidneys, etc.
6. Pathologic type is hepatocellular carcinoma .
7. Confirmation of the presence of VETC vascular pattern by CD34 immunohistochemical staining.

Exclusion Criteria:

1. Pregnant and lactating women.
2. Suffering from a condition that interferes with the absorption, distribution, metabolism, or clearance of the study drug (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, impaired absorption, etc.).
3. A history of gastrointestinal bleeding within the previous 4 weeks or a definite predisposition to gastrointestinal bleeding (e.g., known locally active ulcer lesions, fecal occult blood ++ or more, or gastroscopy if persistent fecal occult blood +) that has not been targeted, or other conditions that may have caused gastrointestinal bleeding (e.g., severe fundoplication/esophageal varices), as determined by the investigator.
4. Active infection.
5. Other significant clinical and laboratory abnormalities that affect the safety evaluation.
6. Inability to follow the study protocol for treatment or follow up as scheduled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | From date of include in this research until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  DFS defined as time to recurrence or death after surgery.

SECONDARY OUTCOMES:
OS | From date of include in this research until the date of death from any cause, whichever came first, assessed up to 60 months
  OS defined as time to death from any cause after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: xiaoping Chen, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code